CLINICAL TRIAL: NCT06269731
Title: Anxiety, Depression and Quality of Life in Thyroid Cancer Patients
Brief Title: Anxiety & Depression in Thyroid Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Mamdouh Mohammed Mahmoud, doctor, Assiut University
Other Study IDs: Thyroid cancer
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Cancer
Keywords: depression; anxiety
MeSH Terms: conditions — Thyroid Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Hamilton depression Rating Scale — also known as the Ham-D is the most widely used clinician-administered depression assessment scale. The original version contains 17 items (HDRS17) pertaining to symptoms of depression experienced over the past week. Although the scale was designed for completion after an unstructured clinical interview, The scale has been translated into a number of languages including French, German, Italian, Thai , Turkish and Arabic version by Mostafa Lotfy.
  Other Names: Hamilton Anxiety Rating Scale; Quality of life Questionnaire; Symptom Checklist-90-Revised

SUMMARY:
1. To identify the prevalence of both anxiety and depression in thyroid cancer patients
2. To assess quality of life in thyroid cancer patients

DETAILED DESCRIPTION:
In recent years, increasing attention has been paid to mental health among cancer patients.

Thyroid cancer is one of the most frequent endocrine neoplasia. It consists of 4 subtypes of papillary thyroid cancer, follicular thyroid cancer, medullary thyroid cancer, and anaplastic thyroid cancer.

Which is usually asymptomatic in the early stages, but symptoms such as neck pain, hoarseness, and dysphagia may occur as the disease progresses. TC is diagnosed by physical examination, analysis of thyroid hormone levels, imaging, and biopsy.

Anxiety and depression are the most common psychological problems in the treatment of cancer patients and are related to the majority of medical diseases and physical symptoms.

Studies have suggested that anxiety and depression are common in patients with thyroid cancer.

Therefore, quality of life which includes psychological, social, and spiritual well-being, has become an important consideration .

These findings highlight the importance of identifying thyroid cancer patients needs to allow better and more adequate care and support.

ELIGIBILITY:
Inclusion Criteria:

1. Age at or more than 18 years old
2. None of the patients had history of other psychiatric illness
3. Both sex
4. Accept to participate in the study

Exclusion Criteria:

1. Age less than 18 years old
2. Previous history of other psychiatric illness
3. substance abuser or dependence
4. Refuse to participate in the study

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: thyroid cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
the prevalence of anxiety in thyroid cancer patients | baseline
  To identify the prevalence of anxiety in thyroid cancer patients by using Hamilton Anxiety Rating Scale
the prevalence of depression in thyroid cancer patients | baseline
  To identify the prevalence of depression in thyroid cancer patients by using Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
assess quality of life in thyroid cancer patients | baseline
  Detect quality of life in patients with thyroid cancer by using Short form 36 Quality of life questionnaire

REFERENCES:
- [Background] Tagay S, Herpertz S, Langkafel M, Erim Y, Bockisch A, Senf W, Gorges R. Health-related Quality of Life, depression and anxiety in thyroid cancer patients. Qual Life Res. 2006 May;15(4):695-703. doi: 10.1007/s11136-005-3689-7. PMID 16688502
- [Background] Dionisi-Vici M, Fantoni M, Botto R, Nervo A, Felicetti F, Rossetto R, Gallo M, Arvat E, Torta R, Leombruni P. Distress, anxiety, depression and unmet needs in thyroid cancer survivors: a longitudinal study. Endocrine. 2021 Dec;74(3):603-610. doi: 10.1007/s12020-021-02786-y. Epub 2021 Jun 18. PMID 34143334
- [Background] Alexander K, Lee SC, Georgiades S, Constantinou C. The "not so good" thyroid cancer: a scoping review on risk factors associated with anxiety, depression and quality of life. J Med Life. 2023 Mar;16(3):348-371. doi: 10.25122/jml-2022-0204. PMID 37168306